CLINICAL TRIAL: NCT01983137
Title: The Efficacy, With Regard to Pain Relief, of Targinact® Treatment for Patients With Severe Pain Compared to Previous Analgesic Treatment; a Non-interventional Study.
Brief Title: A Non-interventional, Observational Study for Targinact® Treatment in Patients With Severe Pain.
Status: Completed | Type: Observational
Sponsor: Mundipharma CVA (Other)
Responsible Party: Sponsor
Other Study IDs: OXN9510
Record Dates: First submitted 2013-04-17; First posted 2013-11-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Severe Pain
Keywords: Chronic pain; Severe pain; oxycodon; naloxon; opioid-induced constipation; opioid; quality of life; laxative; analgesic rescue medication
MeSH Terms: conditions — Pain; Chronic Pain; Opioid-Induced Constipation | interventions — oxycodone naloxone combination; Oxycodone; Naloxone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Targinact® (oxycodone/naloxone)

SUMMARY:
This non-interventional, observational study evaluates the efficacy of Targinact with regard to pain relief in daily clinical practice in Belgium compared to the previous analgesic treatment.

DETAILED DESCRIPTION:
Patients are treated with Targinact® according to daily clinical practice and are monitored during 3 study visits. Parameters assessed are efficacy regarding pain relief, efficacy regarding bowel function, pain relief, use of analgesic rescue medication, bowel function, use of laxatives, safety of Targinact treatment, use of concomitant medication, patient satisfaction and quality of life.

ELIGIBILITY:
Inclusion criteria:

Patients who are to be included in the study, are those who meet all of the following criteria based on the SPC.

1. Male or female patients at least 18 years, or older, with severe pain.
2. Patients with documented history of severe pain treated with WHO step 1, step 2 and/or 3 analgesics with insufficient pain relief and/or unacceptable side effects that require around-the-clock opioid therapy and are likely to benefit from WHO step 3 opioid therapy for the duration of the study.

Exclusion criteria are based on the SPC of Targinact®.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GPs and specialists
Sampling Method: Non-Probability Sample
Enrollment: 1338 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of Targinact® treatment, with regard to pain relief, in patients with severe pain | Up to 140 days
  Efficacy will be evaluated by the physician (7 categories). For the analysis the ordinal scale will be reduced to a binary scale: responder or non-responder. A responder is defined as a patient responding ''slightly better'', ''better'' or ''much better'' at any time during the Targinact®therapy. A non-responder is defined as a patient responding "same", "slightly worse", "worse", "much worse".

SECONDARY OUTCOMES:
Pain NAS score (0-10) will be measured at each visit | Up to 140 days
  The relative changes from baseline at each visit will be used to compare the NAS pain scores during the Targinact® therapy.
Bowel Function Index (BFI) will be recorded at each visit | Up to 140 days
  The Bowel Function Index is the mean value of the 3 single items included in the BFI:1/ Difficulty of bowel movement (0 to 100; 0 = easy/no difficulty, 100 = severe difficulty); 2/ Feeling of incomplete bowel evacuation (0 to 100; 0 = not at all, 100 = very strong); 3/ Judgement of constipation (0 to 100; 0 = not at all, 100 = very strong).
The use of laxative medication (yes/no) per 24 hours will be recorded in the e-CRF | Up to 140 days
  If laxative is used, the physician will document if it's used 1/ continuously, 2/ intermittently or 3/ rarely.
The use of analgesic rescue medication (yes/no) used per day (24 hours) will be recorded | Up to 140 days
Efficacy of Targinact® treatment, with regard to bowel function, will be evaluated by the physician (7 categories) | Up to 140 days
  For the analysis the ordinal scale will be reduced to a binary scale: responder or non-responder. A responder is defined as a patient responding ''slightly better'', ''better'' or ''much better'' at any time during the Targinact® therapy. A non-responder is defined as a patient responding "same", "slightly worse", "worse", "much worse".
The patient satisfaction will be evaluated by patient in 7 categories | Up to 140 days
  much worse, worse, slightly worse, same, slightly better, better, much better.
The patient's quality of life will be evaluated via the EQ-5D questionnaire | Up to 140 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Antwerp (UZA):, Antwerp, Belgium